CLINICAL TRIAL: NCT01783015
Title: A Randomized, Double-blind, Placebo-controlled Study Of The Safety And Efficacy Of Etanercept In Subjects With Rheumatoid Arthritis Who Have Had An Inadequate Response To Adalimumab Or Infliximab Plus Methotrexate
Brief Title: Study of Etanercept in Subjects With Rheumatoid Arthritis Who Have Had an Inadequate Response to Adalimumab or Infliximab Plus Methotrexate
Acronym: SERUM
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was prematurely terminated on June 25, 2014 due to lack of enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1801355; 2012-003644-71 (EudraCT Number)
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Results first posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2015-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; etanercept; methotrexate; infliximab; adalimumab; anti-drug antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): Subjects who are mAb ADA positive
  Interventions: Drug: Etanercept
- Group B (Experimental): Subjects who are mAb ADA negative
  Interventions: Drug: Etanercept
- Group C (Placebo Comparator): Subjects who are mAb ADA positive
  Interventions: Drug: Placebo
- Group D (Placebo Comparator): Subjects who are mAb ADA negative
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg once-weekly
  Arms: Group A
Drug: Etanercept — Etanercept 50 mg once-weekly
  Arms: Group B
Drug: Placebo — Etanercept placebo once-weekly
  Arms: Group C
Drug: Placebo — Etanercept placebo once-weekly
  Arms: Group D

SUMMARY:
The first 12 weeks of this study will compare the efficacy of etanercept 50 mg once-weekly to placebo in subjects with rheumatoid arthritis who have not responded well to infliximab or adalimumab plus methotrexate. This comparison will be performed for all subjects and separately for subjects who are anti-drug antibody positive for one of these medications. From week 12 to week 24, all subjects will receive etanercept 50 mg once-weekly. The effect of anti-drug antibody status on the efficacy of etanercept as well as the safety profile of etanercept in these subjects will also be evaluated throughout the study.

DETAILED DESCRIPTION:
This study was prematurely terminated on June 25, 2014 due to significant and continuing delays in achieving the study B1801355 enrolment target. The decision to stop the study was not driven by any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Met the 1987 ACR Revised Criteria for RA
2. A history of inadequate response to infliximab or adalimumab in combination with methotrexate.
3. A stable dose of oral methotrexate for at least 6 weeks before the baseline visit.

Exclusion Criteria:

1. ACR functional class IV
2. Prior treatment with etanercept; both infliximab and adalimumab; or any immunosuppressive biologic agent other than infliximab or adalimumab.
3. Discontinuation of infliximab or adalimumab for a primary reason other than inadequate efficacy response.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- RK Will Pty Ltd, Victoria Park, Western Australia, Australia
- Cliniques Universitaires Saint-Luc / Service de Rhumatologie, Brussels, Belgium
- Hopital Lapeyronie, Montpellier, France
- Hong Kong (2):
  - Tseung Kwan O Hospital, Tseung Kwan O, New Territories
  - Tseung Kwan O Hospital, Tseung Kwan O, NT
- Israel (2):
  - Bnai Zion Medical Ctr Pharmacy, Haifa
  - Meir Medical Center pharmacy, Kfar Saba
- Russia (4):
  - LLC "Alliance Biomedical - Russian Group", Izhevsk, Russian Federation
  - LLC Research Medical Complex "Your Health" based on City Clinical Hospital #7, Kazan'
  - Scientific Institute of Rheumatology of Russian Academy of Medical Science, Moscow
  - GBOU VPO Moscow State University of Medicine and Dentistry, Moscow
- Spain (4):
  - Hospital de la Santa Creu i San Pau, Barcelona, Barcelona
  - Hospital Regional Universitario Carlos Haya. Hospital Civil, Málaga, Málaga
  - Hospital Regional Universitario Carlos Haya., Málaga, Málaga
  - Hospital Infanta Luisa, Seville

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801355&StudyName=Study%20of%20Etanercept%20in%20Subjects%20with%20Rheumatoid%20Arthritis%20Who%20Have%20Had%20an%20Inadequate%20Response%20to%20Adalimumab%20or%20Infliximab%20Plus%20Methotrex

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this 24 week, multicenter, randomized, double-blind, placebo-controlled (Period 1), 2 period study, a total of 20 participants were screened, out of which 16 participants were randomized. Due to delayed enrollment and an insufficient number of participants, recruitment was terminated.
Pre-assignment Details: Eleven participants were randomly assigned to etanercept [ETN] and 5 participants to placebo in the blinded treatment period. A total of 11 participants (9 ETN treated and 2 placebo treated) completed the blinded treatment period and entered the open label treatment with ETN. One of the 2 placebo treated participants entered the Escape Arm.
Groups:
- Period I - Blinded Treatment - Etanercept: Participants received etanercept 50 mg subcutaneously with oral methotrexate tablets once-weekly.
- Period I - Blinded Treatment - Placebo: Participants received placebo injections with oral methotrexate tablets once-weekly.
- Period 2 - Open Label Treatment: Participants received etanercept 50 mg subcutaneously with oral methotrexate 10 to 25 mg once-weekly.
Period: Blinded Treatment
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Started | 11 | 5 | 0
Treated | 11 | 5 | 0
Completed | 9 | 2 | 0
Not Completed | 2 | 3 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 2 | 0 | 0
Period: Open Label Treatment
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Started | 0 | 0 | 11
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 6
Not completed — Study Terminated by Sponsor | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (13.43) | 54.8 (19.56) | 54.6 (14.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Disease Activity Score Based on a 28 Joint Count (DAS28-C-reactive Protein [CRP]) at Week 12.
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the c-reactive protein (CRP) and Subject General Health Visual Analogue Scale (VAS) assessment (participant rated health assessment with scores ranging 0 to 100; higher scores indicate worse health status).
Time Frame: Baseline, 12 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in the DAS28 at Week 24
Description: DAS28 calculated from the number of SJC and PJC using the 28 joints count, the CRP and and Subject General Health VAS assessment (participant rated health assessment with scores ranging 0 to 100; higher scores indicate worse health status).
Time Frame: Baseline, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With DAS28 <3.2
Description: Number of participants with DAS28 <3.2. A score of < 3.2 implied low disease activity.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With DAS28 <2.6
Description: Number of Participants with DAS28 <2.6. A DAS28 < 2.6 implies remission.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant's assessment of pain; Subject Global Assessment (SGA) of disease activity; Physician Global Assessment (PGA) of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and CRP.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 50% (ACR50) Response
Description: ACR50 response: greater than or equal to (≥) 50 percent (%) improvement in tender or swollen joint counts and ≥ 50% improvement in 3 of the 5 remaining ACR core measures: participant's assessment of pain; SGA of disease activity; PGA of disease activity; subject's assessment of functional disability via a HAQ; and CRP.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 70% (ACR70) Response
Description: ACR70 response: greater than or equal to (≥) 70 percent (%) improvement in tender or swollen joint counts and ≥ 70% improvement in 3 of the 5 remaining ACR core measures: participant's assessment of pain; SGA of disease activity; PGA of disease activity; subject's assessment of functional disability via a HAQ; and CRP.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Number of Participants Achieving American College of Rheumatology 90% (ACR90) Response
Description: ACR90 response: greater than or equal to (≥) 90 percent (%) improvement in tender or swollen joint counts and ≥ 90% improvement in 3 of the 5 remaining ACR core measures: participant's assessment of pain; SGA of disease activity; PGA of disease activity; subject's assessment of functional disability via a HAQ; and CRP.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants Achieving European League Against Rheumatism (EULAR) Good and/or Moderate Response.
Description: The Disease Activity Score Based on 28-joints Count based (DAS28-based) EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 =< 3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to =<5.1 or change from baseline >0.6 to =<1.2 with DAS28 =<5.1; non-responders: change from baseline =< 0.6 or change from baseline >0.6 and =<1.2 with DAS28 >5.1.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Achieving Low Disease Activity or Remission Based on Clinical Disease Activity Index (CDAI)
Description: The CDAI is the numerical sum of 4 outcome parameters: tender joint count (TJC) and SJC based on a 28-joint assessment, SGA and PGA assessed on 0-10 point scale; higher scores=greater affliction due to disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Achieving Low Disease Activity or Remission Based on Simplified Disease Activity Index (SDAI).
Description: The SDAI is the numerical sum of five outcome parameters: TJC) and SJC based on a 28-joint assessment, SGA and PGA assessed on 0-10 point scale; higher scores=greater affliction due to disease activity, and CRP (mg/dL). SDAI total score= 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in CDAI
Description: Change from Baseline in CDAI scores was to be calculated. The CDAI is the numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, SGA and PGA assessed on 0-10 point scale; higher scores=greater affliction due to disease activity. CDAI total score = 0-76. CDAI <= 2.8 indicates disease remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in SDAI.
Description: Change from Baseline in SDAI scores were to be calculated. The SDAI is the numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, SGA and PGA assessed on 0-10 point scale; higher scores=greater affliction due to disease activity, and CRP (mg/dL). SDAI total score= 0-86. SDAI <=3.3 indicates disease remission, >3.4 to 11 = low disease activity, >11 to 26 = moderate disease activity, and >26 = high disease activity.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Number of Tender/Painful Joints
Description: Change from Baseline in the number of tender/painful joints using the 28 joint count including shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints, and knees was to be calculated.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Change From Baseline in Number of Swollen Joints
Description: Change from Baseline in the number of swollen joints including shoulders, elbows, wrists, metacarpophalangeal joints, proximal interphalangeal joints, and knees was to be calculated.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity
Description: Change from Baseline in the PGA scores was to be estimated. The Study Physician estimated the participant's overall disease activity over the last 2 to 3 days using a scale between 0 (no disease activity) and 10 (extreme disease activity).
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in Subject Global Assessment of Disease Activity
Description: Change from Baseline in Subject Global Assessment of Disease Activity was to be estimated. Participants were to assess their overall disease activity over the last 2 to 3 days using a scale between 0 (no disease activity) and 10 (extreme disease activity).
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Subject General Health VAS.
Description: Subject General Health VAS assessment (participant rated health assessment with scores ranging 0 to 100; higher scores indicate worse health status).
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline in Subject Pain
Description: Subject Pain was to be measured on a 0 to 100 mm Visual Analog Scale (VAS), with 0 mm = no pain and 100 mm = most severe pain.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Change From Baseline in CRP
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability and Discomfort Scales (HAQ-DI)
Description: Health Assessment Questionnaire-Disability Index (HAQ-DI): participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Euro Quality of Life (Qol) EQ-5 Dimensions Questionnaire (EQ-5D)
Description: The EuroQol-5 Dimensions (EQ-5D) is a participant-completed questionnaire designed to assess health related quality of life. There are 2 components to the EQ-5D: a Health State Profile and a VAS. For the Health State Profile, participants recorded their level of current health for 5 domains comprising a health profile: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores from the 5 domains may be used to calculate a single index value, also known as a utility score. On the VAS participants were asked to rate their current health on a scale from 0 to 100 mm, where 0 represented the "worst imaginable health state" and 100 represented the "best imaginable health state." In addition to a summary of mean changes, 1 categorical endpoint each based on EQ-5D utility score and 1 based on the VAS were derived and analyzed: EQ-5D utility score improvement ≥0.05 and EQ-5D VAS score >82.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Short Form-36 Health Survey (SF-36)
Description: The 36-Item Short Form Health Survey (SF-36) is widely used 36-item questionnaire that measures general health-related quality of life in the following 8 domains: physical function, role limitations due to physical health, bodily pain, general health perception, vitality, social functioning, role limitation due to emotional problems, and mental health. Scores for the 8 domains range from 0 to 100 where higher scores are better.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Change From Baseline in Patient Acceptable Symptom State (PASS)
Description: The Patient Acceptable Symptom State (PASS) was a participant-completed form in which participants were asked to "Think about all the ways your rheumatoid arthritis (RA) has affected you during the last 48 hours. If you were to remain in the next few months as you were during the last 48 hours, would this be acceptable or unacceptable to you?" The participant indicated a response of either "acceptable" or "unacceptable".
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Change From Baseline in Vectra Disease Activity Levels
Description: The change from Baseline in Vectra disease activity levels was to be estimated. The assessment measures serum protein biomarkers associated with RA. It has a range from 1-100 with lower scores indicating the better outcome.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Vectra disease activity analysis of laboratory samples was not conducted due to study termination.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Positive Etanercept Anti-drug Antibody Status
Description: Blood samples (6 mL) were collected at the baseline, Week 12, and Week 24 visits, or upon early withdrawal, to provide a minimum of 1 mL serum each for ETN ADA and ETN neutralizing antibody analyses. Samples which were positive for ETN anti-drug antibodies were then also tested for ETN neutralizing antibodies.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Positive Etanercept Neutralizing Anti-drug Antibody Status
Description: as for outcome 26
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Due to small sample size, Pfizer did not perform statistical analysis.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the day the first dose of the investigational product was administered up to 28 days after last dose was administered.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Period I - Blinded Treatment - Etanercept | Period I - Blinded Treatment - Placebo | Period 2 - Open Label Treatment
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5 | 0/11
Other Adverse Events (participants affected / at risk) | 5/11 | 3/5 | 4/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period I - Blinded Treatment - Etanercept (N=11) | Period I - Blinded Treatment - Placebo (N=5) | Period 2 - Open Label Treatment (N=11)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 0 | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 0
INJECTION SITE ERYTHEMA (General disorders) | 1 | 0 | 1
INJECTION SITE REACTION (General disorders) | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 1 | 1
TONSILLITIS (Infections and infestations) | 1 | 0 | 1
TOOTH INFECTION (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was prematurely terminated on June 25, 2014. This termination was due to delays in achieving the enrolment target and not due to any safety concerns. No statistical analyses were done since there were a small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.